CLINICAL TRIAL: NCT01788722
Title: Visanne® (Dienogest 2mg) Regulatory Post Marketing Surveillance Study in Korea
Brief Title: Regulatory Post Marketing Surveillance Study in Korea
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16625; VS1310KR (Other: company internal)
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Dienogest (Visanne, BAY86-5258)

INTERVENTIONS:
Drug: Dienogest (Visanne, BAY86-5258) — Patients in daily life clinical practice treatment receiving Visanne (dienogest 2mg) according to indication on the label.

SUMMARY:
The objective of the study is to investigate and collect post marketing data on the safety and efficacy of Visanne at follow-up visit after about 6 months of treatment and - for a subset of patients - at optional long-term follow-up visit after about 1 year of treatment under daily practice treatment conditions in Korean women and to obtain data on drug utilization on treatment for endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Women diagnosed by a physician as having endometriosis
* Women who are prescribed Visanne(dienogest 2mg)for the first time during the study period

Exclusion Criteria:

- All contraindications according to the local marketing authorization have to be considered.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women desiring treatment for endometriosis using Visanne (dienogest 2mg)
Sampling Method: Non-Probability Sample
Enrollment: 3223 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events( AE) and Serious adverse events(SAE) as a measure of safety and tolerability | up to 1 year

SECONDARY OUTCOMES:
Changes of relief of endometriosis-associated pelvic pain (EAPP) will be measured on VAS for total study population | 6 months and 1 year
Evaluation of VAS score changes for sub analysis( In case of VAS score≥ 30mm in initial visit). | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, South Korea